CLINICAL TRIAL: NCT05841888
Title: Implementation of Enhanced Recovery in Women Undergoing Cesarean Delivery Improve Breastfeeding and Maternal Perioperative Outcomes
Brief Title: Implementation of Enhanced Recovery in Women Undergoing Cesarean Delivery
Acronym: ERAS
Status: Completed | Type: Observational
Sponsor: Ali Yavuzcan (Other)
Collaborators: Duygu Yıldız Birden (Unknown); Alper Başbuğ (Unknown); Ali Yavuzcan (Unknown)
Responsible Party: Sponsor-Investigator, Ali Yavuzcan, Head of REI (Reproductive Endocrinology and Infertility), Duzce University
Organization: Duzce University (Other)
Other Study IDs: Ayavuzcan
Record Dates: First submitted 2023-04-04; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: The Aim of Our Study Was to Evaluate the Outcomes in Women Who Implemented the Enhanced Recovery After Surgery Protocol at Delivery by Cesarean Delivery
Keywords: Breastfeeding initation time; cesarean delivery; enhanced recovery after surgery; pain; perioperative outcomes
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: standard perioperative care (SC)
- Group 2: Enhanced Recovery after Surgery (ERAS)

SUMMARY:
Aim: The aim of our study was to evaluate the outcomes in women who implemented the ERAS (Enhanced Recovery after Surgery) protocol at delivery by cesarean delivery(CD).

Methods: The women who underwent CD with ERAS or standard perioperative care (SC) were randomized. In terms of the time to first flatus (TFF), visual pain score (VAS), successful breastfeeding, time of initiation of breastfeeding, time to returning to daily activities, hemoglobin values, postoperative nausea and vomiting, readmission to the hospital, postoperative wound infection, postpartum blues (PB) and the need for blood transfusion were compared between two groups.

DETAILED DESCRIPTION:
Our study was conducted as a prospective study in the Obstetric and Gynecology Department of the Düzce University Faculty of Medicine. The study was initiated after the Düzce University Ethics Committee approval(no: KAEK/2020/239). The study followed the principles set out in the Declaration of Helsinki. Pregnant women aged ≥18 years and ≥37 weeks of gestational age who were admitted to our hospital between November 2020 and February 2021 were included in the study. Pregnant women who underwent CD with an indication for emergency cesarean (pregnancy complications such as preeclampsia, placenta previa, detached placenta, fetal distress, infection, disease causing systemic morbidity, or intestinal adhesions secondary to previous operations) were excluded. In addition, pregnant women with any substance addiction and those who did not give informed consent were excluded from the study. Women who did not comply with the study protocols during were not included. Informed consent was obtained from all pregnant women before starting the study. Women who accepted to participate in the study and met the criteria were given the ERAS and control group protocol cards without being shown, upside down, and patients who would or would not receive the ERAS protocol were randomized accordingly. Age, body mass index (BMI), gravidy, parity, gestational age, indication, hemogram value, anesthesia method, presence of comorbidities, and contact information were recorded.

Women who underwent CD and received standard perioperative care (SC) constituted the control group.15 Patients in the SC group who were hospitalized for CD were discontinued from oral water intake and nutrition preoperatively at 00:00 the night before CD. Pethidine hydrochloride was administered as an opioid in addition to postoperative oral paracetamol and parenteral diclofenac sodium after surgery. The bladder catheter was withdrawn at the 6 th postoperative hour, and out-of-bed mobilization was started then. Oral feeding was started after first flatus. Dressings were applied in the morning on the 1st and 2nd postoperative day.

Pregnant women to whom the ERAS protocol would be implemented were given detailed information by explaining the preoperative, intraoperative, and postoperative ERAS elements. They signed the informed consent forms. The study group was formed with patients who received the ERAS protocol. The ERAS Practice Guideline in CD for the pre-operative, intra-operative and post-operative care were implamented.16-18 The women in ERAS group was not be encouraged to drink clear liquids until 2 hour (h) before surgery, to eat a light meal 6 h before surgery or to receive oral carbohydrate supplementation 2 h before CD since the anesthesia department of our hospital did not approve. We could not given antacids and histamine H2 receptor as premedication to women in ERAS group. All of the subjects implemented or not in both ERAS and SC groups were summarized in Table 1. Perioperative information and implementation of ERAS protocol items were checked and recorded in the ERAS protocol checklist. After discharge, patients were called from the contact addresses they provided to check their status and get information and were called to the outpatient clinic within 2 weeks after discharge.

Postoperative pain was calculated with the visual pain score (Visual Analog Scale, VAS) in all patients included in our study. All patients in SC group and in the ERAS protocol group were asked to place a line between 0 and 10 on a horizontal line describing their pain status. The mildest pain represented as 0 and 10 represented the most severe pain.19 The time of first flatulence (TFF)20 and the time of first breastfeeding were recorded as hours. Women were asked when they were able to do things such as eating, walking, and taking care of their baby without assistance and feeling comfortable. The time to return to daily activities is indicated in days. Patients who re-admitted to the hospital within 30 days were considered as readmission.20 The preoperative Hb and the postoperative Hb level (ΔHb) were calculated as gr/dl. It has been accepted that successful breastfeeding is achieved in newborns who are given only breast milk in the appropriate position without formula or additional food.21 The Coronavirus disease (COVID-19) pandemic has been shown to induce a desire for early discharge in all patients after CD.22-23 In our study, an objective evaluation of length of hospital stay could not be made since the discharge times of the patients were affected by COVID-19 pandemic.

The study results were reported in accordance with the CONSORT guideline.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* aged ≥18 years
* ≥37 weeks of gestational age
* admitted to our hospital.

Exclusion Criteria:

* Pregnant women who underwent CD with an indication for emergency cesarean (pregnancy complications such
* preeclampsia,
* placenta previa,
* detached placenta,
* fetal distress, infection,
* disease causing systemic morbidity,
* intestinal adhesions secondary to previous operations) .
* pregnant women with any substance addiction
* those who did not give informed consent were excluded from the study.
* Women who did not comply with the study protocols during were not included.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women aged ≥18 years and ≥37 weeks of gestational age who were admitted to our hospital.
Study Population: Pregnant women aged ≥18 years and ≥37 weeks of gestational age who were admitted to our hospital.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 30 day
  Visual Analogue Scale
Time to first flatus | 30 day
  hour
time to returning to daily activities | 30 day
  day
ΔHb | 30 day
  gr/dl

SECONDARY OUTCOMES:
the breastfeeding initiation time | 30 day
  hour
Successful breastfeeding | 30 day
  newborns who are given only breast milk in the appropriate position without formula or additional food

CONTACTS AND LOCATIONS:
Overall Officials: Ali S Yavuzcan, PhD, Study Director — Duzce University
Locations (1):
- Ali Yavuzcan, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No